CLINICAL TRIAL: NCT00804206
Title: Phase 4 Comparison of the Effects of Bevacizumab Before vs After Pattern Panretinal Photocoagulation
Brief Title: Comparison of the Effects of Bevacizumab Before vs After Pattern Panretinal Photocoagulation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-040
Record Dates: First submitted 2008-12-03; First posted 2008-12-08 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Macular Edema
Keywords: Intravitreal injection of Bevacizumab; Visual acuity; central retinal thickness; color studies, Farnsworth-Munsell; electroretinogram studies
MeSH Terms: conditions — Macular Edema | interventions — Bevacizumab

ARMS (2):
- Group A (Experimental): Bevacizumab before panretinal photocoagulation.
  Interventions: Drug: bevacizumab
- Group B (Experimental): Bevacizumab after panretinal photocoagulation
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab — Intravitreal bevacizumab before panretinal photocoagulation
  Arms: Group A
Drug: bevacizumab — Intravitreal Bevacizumab after panretinal photocoagulation
  Arms: Group B

SUMMARY:
Compare the effect of an intravitreal injection of bevacizumab previous or posterior of panretinal laser photocoagulation (PRLP) with a pattern laser; to prevent and reduce diabetic macular edema (DME) in patients with proliferative diabetic retinopathy (PDR) with DME.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proliferative diabetic retinopathy
* patients with macular edema

Exclusion Criteria:

* patients with previous treatments
* patients with ocular surgeries

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Central macular thickness | baseline, 10 days, 52 days, 85 days

SECONDARY OUTCOMES:
Best corrected visual acuity | baseline, 10 days, 52 days, 85 days

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación para Evitar la Ceguera en México, México, Mexico